CLINICAL TRIAL: NCT04470895
Title: Impact of Drugs on the Risk of Falls in the Fracture Department of the Paris Saint-Joseph
Brief Title: Impact of Drugs on the Risk of Falls in the Fracture Department of the Paris Saint-Joseph Hospital Group
Status: Withdrawn | Type: Observational
Why Stopped: The PI chose not to start the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MEDI-CHUTE
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Fracture; Fall
Keywords: elderly; ageing
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual falling patients: a group enrolling the patients who completed the inclusive criteria and have had at least one fall in the last 12 months in addition to the possible fall causing the index fracture.
  These patients must answer positively the following question "Have you fallen in the last 12 months, regardless of the current fracture"?
  Interventions: Diagnostic Test: Failure Track patients analysis
- Unusual falling patients: a group enrolling the patients who also completed the inclusive criteria, but are defined as "unsual falling patients". These patients must answer negatively the following question: "Have you fallen in the last 12 months, regardless of the current fracture"?
  Interventions: Diagnostic Test: Failure Track patients analysis

INTERVENTIONS:
Diagnostic Test: Failure Track patients analysis — The nurse coordinator of the Fracture Track first comes to give the patient a written information note. She answers the patient's questions and obtains his or her non-opposition. The patient must be given sufficient time for reflection to make his decision in order to participate in the study. His non opposition will be traced in the computerized medical record. Each enrolling patient in the study can simultaneously participate in another research. There is no exclusion period in the protocol.
  Once the patient is included, a semi-directed interview is conducted. The name of the patient's usual pharmacy will be collected. Data from the computerised medical record concerning the patient's stay are also analysed.
  The patient's usual pharmacy or the nurse in charge of the patient will then be questioned in order to carry out a drug reconciliation interview.

SUMMARY:
Falls of the elderly are a public health problem that have been neglected for too long. The experience of a fall makes the elderly person vulnerable, even in the absence of traumatic consequences, and can sometimes be a reason for institutionalization. These falls are frequent and have many repercussions on the autonomy of seniors. According to data from the National Institute for Prevention and Health Education (INPES), falls are the leading cause of accidental death among people over 65 years of age. They cause approximately 8,500 deaths per year. After the age of 65, one person in three falls at least once a year. They account for 10% of the reasons for consultation and 12% of hospitalizations in geriatric settings among the elderly. The risk increases with age because 80% of people over 85 years of age fall at least once a year. 20 to 30% of people over 65 have a loss or decrease in autonomy after a fall. The risk of another fall is twenty times higher after a first fall and the risk of death increases especially in the year following the fall. This is of major importance because falls are responsible for the majority of fractures in the elderly, especially femoral neck fractures. The cost of falls among the elderly is significant and estimated at 2 billion euros for communities.

DETAILED DESCRIPTION:
The causes of falls are multiple and the imputability of medication is often mentioned. In fact, physiological or pathological ageing, which often justifies an intensification of drug use, leads to polymedication, which is recognised as a risk factor for falls in the elderly and generates dosage regimens that are most often complex and which are a source of drug over- or under-dosage. Thus, a large number of treatments increase the risk of drug interactions, particularly of a pharmacokinetic nature, which may lead to drug overdoses, while poor compliance with prescriptions may lead to underdoses. The main classes of drugs currently attributed to the risk of falls are psychotropic drugs, sleeping pills and tranquillizers, antidepressants, cardiovascular drugs, antiepileptics, hypoglycemic drugs and drugs that cause orthostatic hypotension such as antihypertensives.

Screening for risk factors for falls is an important step in management. The recommendations drawn up by the Société Française de Documentation et de Recherche en Médecine Générale (SFDRMG), in partnership with the Haute Autorité de Santé (HAS), suggest specifying the relevant interventions, both medicinal and non-pharmaceutical, to avoid an initial fall (indications, necessary means, interactions between the interveners).

Osteoporosis is a diffuse skeletal disease characterized by low bone mass and deterioration of the micro-architecture of bone tissue, responsible for an increased risk of fracture. The prevention of osteoporotic fractures is essential and involves screening and treatment of osteoporosis but also the prevention of falls. New care pathways have been developed in recent years, in particular the Fractures Liaisons Services to improve the management of this pathology.

Fracture Pathways (in English: Fractures Liaisons Services: FLS), so called because of the need for a link between the services concerned by this pathology (emergency, orthopaedic surgery, rheumatology, sometimes geriatrics), aim to identify, screen and, if necessary, treat patients with osteoporosis.

Within the Paris Saint-Joseph Hospital Group (GhSPJ), the OPTIPOST study (OPTImisation de la Prise en Charge de l'OSTéoporose chez des sujets de plus de 45 ans) highlighted the benefits of "reinforced" management of patients with osteoporotic fractures of the upper end of the femur (ESF) or the lower end of the radius (EIR) via a specific organisation coordinated by an IDE between 2014 and 2015.

This is why, following these results, and in the continuity of OPTIPOST, a Fracture Track has been set up at the GhPSJ. This is a new organisation dedicated to the management of fractured osteoporosis, independent of OPTIPOST, based on the census and follow-up of patients aged 45 to 95 years old admitted to the emergency reception service (UAS) for any kind of osteoporotic fracture. The main objective of this approach is the management of fractured osteoporosis. Patients included in this line are counted by the nurse coordinator on D0 and are questioned by telephone within 2 months following the fracture to ensure that the osteoporosis is being managed.

Currently, the Fracture Track does not take into account the risk factors for falls in osteoporotic fractured patients, in particular the risk of falls due to medication, hence the aim of this work.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 45 and 95
* French-speaking
* Patient included in the GhPSJ fracture track, taking at least one long-term prescription medication and hospitalized in a GhPSJ department or in Léopold Bellan.

Exclusion Criteria:

* Patient objecting to participation in the study
* Patient who has recently moved or medical nomadism making it impossible to reconcile medication with a pharmacy
* Patient not hospitalized or transferred to a hospital other than the GhPSJ or Léopold Bellan at the time of the fracture
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under the safeguard of justice.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study involving patients aged between 45 and 95 years, who is affiliated to the fracture track and has taken various types of medications after a fall that has occurred in the last 12 months
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Impact of drugs on Fracture Track Patients | July, 2020
  The research aims at determining the impact of drug intake (number and type of drugs) on the occurrence of falls in patients hospitalized for an osteoporotic fracture.

SECONDARY OUTCOMES:
Frequency of falls on Fracture Track patients. | July, 2020
  The research also aims at determining the frequency of fall in fracture Tracks patient and the frequency of self medication, as well as the possible therapeutics changes made by the caregivers following the occurrence of the fall on criteria such as the prescription changes, the drug addition/ deletions molecule changes... It will also evaluate the influence of age/ age range on medication use and the occurrence of falls and establish an algorithm for managing the drug risk of falling in the fracture track.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Chute sur la personne âgée: causes, conséquences et prévention — https://www.silvereco.fr/chute-de-la-personne-agee-causes-consequences-et-prevention/3187245
- See also: Médicaments et chutes [Internet] — http://www.iugm.qc.ca/sante-aines/infochute/chute-corps/chute-corps-medicament.html